CLINICAL TRIAL: NCT05498077
Title: Immediate Effects of a 10-minute Body Scan Meditation on People Who Has Central Sensitization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Therapeutic Neuroscience Research Group (Network)
Collaborators: Rockhurst University (Other); Evidence In Motion (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSFMcConahay
Record Dates: First submitted 2022-08-08; First posted 2022-08-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Chronic Pain
Keywords: Central Sensitization; Meditation
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Case series
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 10 minute body scan meditation (Experimental): Participants will be taken through a 10 minute body scan meditation by a physical therapist
  Interventions: Procedure: Body scan meditation

INTERVENTIONS:
Procedure: Body scan meditation — Subject is placed through a brief body scan meditation to determine whether this intervention affects a person's pain experience

SUMMARY:
For patients with chronic pain, how does a 10 minute guided body scan meditation affect pressure pain threshold and extent of pain on a body diagram?

DETAILED DESCRIPTION:
Patients who present with central sensitization in physical therapy will go through a 10 minute body scan meditation. If patient meets criteria then they will fill out pre-intervention measures including hand dominance, gender identity, duration of pain, work status, pain body diagram, current pain level, previous medication and a neck disability index or an oswestry disability index.

Subject will then be asked what position they feel most comfortable to be led through this body scan meditation.

After the meditation, the participant will fill out another pain body diagram, current pain level, global rating of change and pain pressure threshold.

At this point the study is over and the subject will return to their physical therapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are from a convenience sample of patients seeking physical therapy care from a physician referral or direct-access to a privately owned physical therapy clinic English speaking
* Central Sensitization Inventory > 40
* Subject complains of disproportionate non mechanical unpredictable pattern of pain provocation in response to multiple non-specific aggravating/easing factors
* Pain disproportionate to the nature and extent of injury or pathology
* Strong association with maladaptive beliefs and pain behaviors
* Diffuse, nonanatomic areas of pain and tenderness on palpation

Exclusion Criteria:

* Does not meet the criteria above

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Global Rating of Change | Immediately After intervention
  This is a form the subject fills out rating their overall pain experience after an intervention. The scale is from -7 (Significantly worse to +7 Significantly better) and measures the amount of change the person feels they have experienced.
Pain pressure Threshold | Immediately Before and immediately after intervention
  This is a pressure algometer the measures the sensitivity of an area on the body to direct pressure. It measures the amount of pressure that is applied to the subject's body. The clinician will apply pressure to the subject's skin at the tibialis anterior, lumbar paraspinals and upper trapezius muscles on the dominant hand side. The clinician will ask the subject "I want you to tell me the moment the sensation changes from pressure to discomfort and say "STOP". That is the reading/measurement the clinician will take. The outcome is assessing a change in pressure discomfort before the meditation and immediately after the meditation.
Neck Disability Index | Immediately Before the intervention
  This is a questionnaire to measure the amount of disability the subject perceives due to their neck pain.
Oswestry Disability Index | Immediately Before the intervention
  This is a questionnaire to measure the amount of disability the subject perceives due to their back pain
Pain Body Diagram | Immediately Before the intervention and immediately after intervention
  This is an body image drawing. The subject colors in the area on the image of where they are experiencing pain. This outcome is assessing the location and extent of the area of pain in the body and how it changes with the intervention. The way this is assessed is by dividing the body image drawing into a grid. The body pain diagram consists of an outline of the entire body from anterior and posterior views. An overlay is created dividing the body pain diagram into 45 anatomical regions The overlay is placed over the body pain diagram, and the examiner recorded a score of 1 if pain is indicated and 0 if no pain is indicated in each of the 45 regions. Pain is considered present if any portion of the region was shaded, no matter how small.
Numeric Pain Rating Scale | Immediately Before the intervention and immediately after intervention
  This is a scale assessing the subjects pain. It is a scale from 0 (no pain) to 10 (being the most severe pain). The subject will be assessed if their pain rating changed from before the intervention to after the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Whole Body Health Physical Therapy, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No